CLINICAL TRIAL: NCT05875649
Title: A Multicenter Prospective Cohort Study Study of CLAG Regimen in Acute Myeloid Leukemia Patients With First-induction Failure
Acronym: CLAG
Status: Not yet recruiting | Type: Observational
Sponsor: Nanfang Hospital, Southern Medical University (Other)
Responsible Party: Sponsor
Other Study IDs: NEFC-2023-162
Record Dates: First submitted 2023-05-16; First posted 2023-05-25 (Actual); Last update posted 2023-07-05 (Actual); Status verified 2023-07

CONDITIONS: AML
Keywords: CLAG; acute myeloid leukemia; First-induction failure
MeSH Terms: conditions — Leukemia, Myeloid, Acute

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 24 Months
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Group: Acute myeloid leukemia patients with first-induction failure
  Interventions: Combination Product: CLAG

INTERVENTIONS:
Combination Product: CLAG — Acute myeloid leukemia patients are re-induced by CLAG Regimen after first-induction failure

SUMMARY:
Most of patients with acute myeloid leukemia achieved complete remission (CR) after primary induction chemotherapy, there were 20-30% patients without CR after first-induction. It was uncertain how to treat these patients. It was investigated in our study that these patients were re-induced with CLAG Regimen. The CR ratio, overall survival (OS) and relapsed-free survival (RFS) was statistically analysed in these patients.

ELIGIBILITY:
Inclusion Criteria:

* Acute myeloid leukemia patients with first-induction failure

Exclusion Criteria:

* Acute myeloid leukemia patients with serious infection and organ dysfunction.

Ages: 14 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Acute myeloid leukemia patients don't achieve CR after first-induction chemotherapy.
Sampling Method: Non-Probability Sample
Enrollment: 137 (Estimated)
Dates: Start 2023-07-02 (Estimated); Primary Completion 2027-08-20 (Estimated); Study Completion 2027-12-20 (Estimated)

PRIMARY OUTCOMES:
Study of CLAG Regimen in Acute Myeloid Leukemia Patients With First-induction failure | 6 months
  CLAG Regimen improves CR rate in acute myeloid leukemia patients with first-induction failure

CONTACTS AND LOCATIONS:
Overall Officials: Xuejie Jiang, Doctor, Study Chair — Nanfang Hospital, Southern Medical University
Locations (1):
- Nanfang Hospital of Southern Medical University, Guanzhou, Guangdong, China

IPD SHARING:
Plan to Share IPD: No
CLAG Regimen is used to re-induce acute myeloid leukemia patients after first-induction failure